CLINICAL TRIAL: NCT06016907
Title: A Pilot Randomized Controlled Trial of Stepped vs Stratified Care for Pediatric Anxiety Disorders
Brief Title: Stepped vs Stratified Care for Pediatric Anxiety Disorders
Acronym: PMAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-07219-01
Record Dates: First submitted 2023-08-16; First posted 2023-08-30 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders; Children; Adolescents; Cognitive behavioral therapy; RCT; Care pathway; Stepped care; Stratified care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A pilot, single-blind, parallel-group (2 groups), randomized controlled trial for children and adolescents with anxiety disorders. Participants will be randomized at a 1:1 ratio to one out of two care pathways: stepped care and stratified care. Each care pathway consists of up to two courses of treatment.
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting follow-up assessments (referred to as POST-1 and POST-2) will be blind to treatment allocation. At each follow-up assessment, participants will be reminded by their assessor to not reveal their study allocation. To measure blinding integrity, all assessors will record whether the participants inadvertently revealed their group allocation, and subsequently guess each participant's treatment allocation at each assessment point and motivate their choice. If the treatment allocation is accidentally revealed, the revelation part will be cut out of the Pediatric Anxiety Rating Scale audio recording and a new blind assessor will listen to the audio recording and conduct the rating that will be used in the trial. Subsequent assessments for that participant will then be conducted by someone different than the unblinded assessor. The primary analysis will be performed after the study's final participant has finished his/her POST-2 assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped care (Other): Participants will receive up to two courses of treatment. All participants in stepped care will receive internet-delivered cognitive behavioral therapy (ICBT) in the first course (A). Participants with an insufficient treatment response will then be offered in-person cognitive behavioral therapy (CBT) in the second course (B). Even if participants are offered treatment in course B, participants are free to decline this offer, and will instead only be invited to the remaining outcome assessments.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy (ICBT); Behavioral: In-person cognitive behavioral therapy (CBT)
- Stratified care (Other): Participants will receive up to two courses of treatment. In stratified care, in treatment course A, the investigators aim to offer around half of the participants ICBT and the other half in-person CBT (based on their risk of non-response). All participants in stratified care who do not sufficiently respond to treatment in course A will be offered personalized in-person CBT in course B. Even if participants are offered treatment in course B, participants are free to decline this offer, and will instead only be invited to the remaining outcome assessments.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy (ICBT); Behavioral: In-person cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy (ICBT) — Cognitive behavioral therapy (CBT) delivered through an internet platform with therapist support.
Behavioral: In-person cognitive behavioral therapy (CBT) — Cognitive behavioral therapy (CBT) delivered in-person at a clinic by a therapist.

SUMMARY:
The purpose of this trial is to evaluate the feasibility, acceptability, and safety of two care pathways (including internet-delivered cognitive behavioral therapy [CBT] and/or in-person CBT) for children and adolescents with anxiety disorders.

DETAILED DESCRIPTION:
Introduction: Anxiety disorders are a major contributor to disability in children and adolescents. Cognitive behavioral therapy (CBT), delivered both in-person and by the internet (ICBT), is efficacious, but how to best organize the care pathway to increase access and benefit is unclear.

Methods: With the aim to conduct a fully powered randomized controlled trial, the present study is a randomized controlled, single-blind, pilot study where 50 youth with anxiety disorders and their caregivers will be randomized (1:1) to stepped care or stratified care. Stepped and stratified care are two competing service delivery models which include evidence-based interventions but differ regarding the timing and staging of interventions.

In the stepped care arm, all participants will begin with 12 modules of ICBT delivered over 12 weeks. Participants with an insufficient response will then be offered 12-weeks of personalized in-person CBT. In the stratified care arm, the investigators aim to offer about half of the participants ICBT and the other half in-person CBT, with this selection being based on a risk score algorithm that integrates known predictors of non-response to treatment.

Mirroring the structure in stepped care, all non-responders in stratified care (both those who started with ICBT and in-person CBT) will be offered an additional 12-week course of in-person CBT. The ICBT and in-person CBT interventions will be identical in treatment length, but will differ in the delivery of treatment, utilizing the possibility of increased personalization and therapist-involvement in in-person CBT.

The objectives of the pilot study are to examine feasibility, acceptability, and safety of study procedures, precision of the risk score algorithm, and statistical properties of outcome measures. The feasibility, acceptability, and safety objectives are operationalized in detail in the full study protocol published at the Open Science Framework (OSF; see link in the References-section at the bottom of this record).

Data will be collected at baseline, post-allocation (week 1), weekly during treatment course A (week 2-13), after treatment course A (POST-1; time window for data collection between week 14-17), weekly during treatment course B (if applicable, week 18-29), and after treatment course B (POST-2; time window for data collection between week 30-33). POST-2 is the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

1. 8 to <18 years of age.
2. A principal Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) anxiety disorder of social anxiety disorder, generalized anxiety disorder, panic disorder, separation anxiety disorder, specific phobia, or agoraphobia.
3. A Clinical Global Impression Scale - Severity (CGI-S) score >3 in relation to severity of all anxiety symptoms.
4. Child and caregiver able to read, write and communicate in Swedish.
5. An available caregiver who can support the child in treatment.
6. Access to the internet.
7. Ability to attend treatment sessions at the clinic.

Exclusion Criteria:

1. Principal DSM-5-TR anxiety disorder of specific phobia concerning the domain of blood-injection-injury (due to the ICBT program not including relevant information on applied-tension techniques to avoid fainting during exposure exercises).
2. Established or suspected intellectual disability.
3. Another mental disorder in more immediate need of management than an anxiety disorder (e.g., schizophrenia spectrum and other psychotic disorders, bipolar disorder, anorexia nervosa, substance use disorders).
4. Social/familial/educational difficulties in more immediate need of management than an anxiety disorder.
5. Ongoing psychological treatment for an anxiety disorder.
6. Initiation or adjustment of any psychotropic medication for anxiety (i.e., selective serotonin reuptake inhibitors, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitor or antipsychotics) within 8 weeks prior to assessment.
7. Immediate risk to self or others that require urgent attention, such as suicidality.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess anxiety severity. Clinician-rated. Primary clinical outcome of the study. The scale yields a score of 0 to 35, with higher scores indicating more severe anxiety.

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess anxiety disorders and psychiatric comorbidity at baseline and anxiety disorders and major depression at follow-ups. Clinician-rated.
Clinical Global Impression Scale - Severity (CGI-S) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess overall anxiety severity. Clinician-rated. Ratings are reported on a seven-graded scale from 1 ("Normal, not at all ill") to 7 ("Among the most extremely ill patients").
Clinical Global Impression Scale - Improvement (CGI-I) | POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess level of improvement compared to admission. Clinician-rated. This single item scale ranges from 1 ("Very much improved") to 7 ("Very much worse").
Children's Global Assessment Scale (CGAS) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess global impairment. Clinician-rated. The CGAS is a single item scale that ranges from 1 to 100, with a higher value indicating better functioning.
Number of participants with concomitant interventions | POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess potential other treatments during the study period. Clinician-rated.
Measure of accidental unmasking | POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess the number of occasions where outcome assessors are accidentally unmasked to group allocation.
Guess of group allocation | POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess the percentage of correctly guessed group allocation from masked outcome assessors.
Experiences of participating in the study | POST-2 (week 30-33).
  A semi-structured interview conducted by a non-masked study coordinator covering (i) burden of participation, (ii) experiences of interventions, (iii) understandability of measures/interviews, and (iv) missing content in measures/interviews. Clinician-rated.
Interviews with participants about treatment | POST-1 (week 14-17) or POST-2 (week 30-33).
  A semi-structured interview conducted by a non-masked researchers who is not otherwise involved in the study covering topics about treatment content, treatment timing, degree of therapist contact, caregiver collaboration and personal effort/motivation as well as themes important to the child/adolescent. Clinician-rated.
Revised Child Anxiety and Depression Scale - Child version (RCADS-C) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess anxiety symptoms. Child/adolescent-reported. The RCADS version used in the present study is the 47-item version which ranges from 0 to 141 points, with higher scores indicating more severe internalizing symptoms.
Child Anxiety Life Interference Scale - Revised - Child version (CALIS-R-C) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess life interference and impairment associated with childhood anxiety. The scale ranges from 0 to 36 points, with higher scores indicating higher interference and impairment.Child/adolescent-reported.
Deliberate Self-harm Inventory - Youth version (DSHI-Y) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess self-harm. Child/adolescent-reported.
Ill temper scale of the Inventory of Depression and Anxiety Symptoms II - Child version (IDAS-II-C) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess irritability. Child/adolescent-reported. The scale ranges from 0 to 20 points, with higher scores indicating greater anger.
Child Health Utility 9D (CHU9D) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess health-related quality of life. Child/adolescent-reported. The scale ranges from 9 to 45 points, with higher scores indicating worse quality of life.
Systematic Clinical Outcome and Routine Evaluation-15 - Child version (SCORE-15-C) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess family functioning. Child/adolescent-reported. The scale ranges from 15 to 75, with a lower score indicating higher family functioning.
Need for treatment - Child version | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess need of treatment for anxiety symptoms. Child/adolescent-reported. This single item scale ranges from 1 to 5 points, with higher scores indicating a higher need for treatment.
Client Satisfaction Questionnaire - Child version (CSQ-8-C) | POST-1 (week 14-17); POST-2 (week 30-33; only if a second round of treatment is initiated).
  Used to assess treatment satisfaction. Child/adolescent-reported. The scale ranges from 9 to 36 points, with higher scores indicating greater satisfaction.
Adverse events questionnaire - Child version (AEQ-C) | Every third week during week 2-13 and 18-29 (the latter applies only if a second round of treatment is initiated).
  Used to assess adverse events/effects. Child/adolescent-reported. The scale consists of 22 yes/no items (score range 0-22 points) with higher scores indicating more present adverse events. For each adverse event that is present, there is also a rating of whether the adverse event is thought to be related to the provided treatment (yes or no).
Working alliance - Child version | Every third week during weeks 2-13 and 18-29 (the latter applies only if a second round of treatment is initiated).
  Used to assess the participant's perceived working alliance with their therapist. Child/adolescent-reported. The scale ranges from 0 to 36 points, with higher scores indicating better working alliance.
Revised Child Anxiety and Depression Scale - Parent version (RCADS-P) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess anxiety symptoms. Caregiver-reported. The RCADS version used in the present study is the 47-item version which ranges from 0 to 141 points, with higher scores indicating more severe internalizing symptoms.
Child Anxiety Life Interference Scale - Revised - Parent version (CALIS-R-P) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess life interference and impairment associated with childhood anxiety. Caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating higher interference and impairment.
Systematic Clinical Outcome and Routine Evaluation-15 - Parent version (SCORE-15-P) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess family functioning. Caregiver-reported. The scale ranges from 15 to 75, with a lower score indicating higher family functioning.
Ill temper scale of the Inventory of Depression and Anxiety Symptoms II - Parent version (IDAS-II-P) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess irritability. Caregiver-reported. The scale ranges from 0 to 20 points, with higher scores indicating greater anger.
Need for treatment - Parent version | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess need of treatment for anxiety symptoms. Caregiver-reported. This single item scale ranges from 1 to 5 points, with higher scores indicating a higher need for treatment.
The Treatment Inventory of Costs in Patients With Psychiatric Disorders (TIC-P) | Baseline; POST-1 (week 14-17); POST-2 (week 30-33).
  Used to assess healthcare and other societal resource use for both children and caregivers. Caregiver-reported.
Client Satisfaction Questionnaire - Parent version (CSQ-8-P) | POST-1 (week 14-17); POST-2 (week 30-33; only if a second round of treatment is initiated).
  Used to assess treatment satisfaction. Caregiver-reported. The scale ranges from 9 to 36 points, with higher scores indicating greater satisfaction.
Adverse events questionnaire - Parent version (AEQ-P) | Every third week during week 2-13 and 18-29 (the latter applies only if a second round of treatment is initiated).
  Used to assess adverse events/effects. Parent-reported. The scale consists of 22 yes/no items (score range 0-22 points) with higher scores indicating more present adverse events. For each adverse event that is present, there is also a rating of whether the adverse event is thought to be related to the provided treatment (yes or no).
Working alliance - Parent version | Every third week during weeks 2-13 and 18-29 (the latter applies only if a second round of treatment is initiated).
  Used to assess the caregiver's perceived working alliance with their therapist. Caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating better working alliance.
Behavioral, Emotional, and Social Skills Inventory (BESSI) | Week 1; POST-2 (week 30-33).
  Used to assess emotional resilience and self-management. Child/adolescent and caregiver-reported. The scale consists of 102 items, each rated from 1 to 5 points, and scores are presented as averages on six different combinations of items, referred to as "Skill domains".
The PROMIS peer relationships short form (PR-SF) | Week 1; POST-2 (week 30-33).
  Used to assess peer relationships. Child/adolescent-reported. The scale ranges from 8 to 40 points, with higher scores indicating greater peer relationships.
Avoidance and Fusion Questionnaire for Youth (AFQ-Y8) | Week 1; POST-2 (week 30-33).
  Used to assess psychological inflexibility. Child/adolescent-reported. The scale ranges from 0 to 32 points, with higher scores indicating greater psychological inflexibility.
The Cognitive-attentional Syndrome Questionnaire (CAS-1) | Week 1; POST-2 (week 30-33).
  Used to assess dysfunctional metacognitive beliefs. Child/adolescent-reported. The questionnaire consists of four domains. Each item of the three first domains is scored on a 0-8 point scale. Each item of the fourth domain is score on 0-100 scale. Higher scores indicates more dysfunctional metacognitive beliefs.
Hierarchical Personality Inventory for Children (HiPIC-30) | Week 1.
  Used to assess personality traits. Child/adolescent and caregiver-reported. The questionnaire collects data on five personality domains. Each of the 30 items range from 1 to 5 points. Higher scores indicates greater indication of the personality domain in question.
Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) | Week 1; POST-2 (week 30-33).
  Used to assess attention difficulties, hyperactivity, impulsivity, and oppositional symptoms. Caregiver-reported. Each item is scored from 0 to 3 points. The item scores are then summarized in domains: inattention (items 1-9), hyperactivity-impulsivity (items 11-19) and oppositional (items 21-28). Items 10, 20 and 29 are not included in any of the domains. Higher scores indicate greater attention difficulties, hyperactivity, impulsivity, and oppositional symptoms.
Autism Phenotype Scale (APS) | Week 1; POST-2 (week 30-33).
  Used to assess core autism traits. Child/adolescent and caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating greater autism traits.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Region Skane and Lund University
Locations (1):
- Child and Adolescent Mental Health Services, Region Skane, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The data are pseudonymized according to national (Swedish) and European Union legislation and cannot be anonymised and published in an open repository. Participants in the study consent for their data to be shared with other international researchers for research purposes. The data can be made available upon reasonable request on a case-by-case basis according to the current legislation and ethical permits.

REFERENCES:
- See also: All full study protocol versions are available at this open repository. — https://osf.io/k6j7n/